CLINICAL TRIAL: NCT03907813
Title: The Effect of Local Infiltration of Liposomal Bupivacaine on Opioid Consumption at Time of Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine After Cesarean Delivery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: change in design
Sponsor: Wright State University (Other)
Responsible Party: Principal Investigator, Marilyn J Kindig, D.O., Assistant Professor, Wright State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kindig-Williams-001
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- liposomal bupivacaine infiltration (Experimental): Local infiltration of all wound layers with liposomal bupivacaine (Exparel(R)) 20 ml diluted with 70 ml of normal saline to 90 ml for patient with a BMI of 39 and under. If BMI is 40 or more the 20 ml of liposomal bupivicaine will be diluted to 150 ml by adding 130 ml of normal saline
  Interventions: Drug: Exparel
- Saline infiltration (Placebo Comparator): Local infiltration of all wound layers with saline, using to match the amount. The amount of total fluid is divided into 4 and instilled with 1-2 ml at a time in between fascial layers after fascial closure. Each 1/4 will be instilled laterally (2) and on each side of the incision(2)- extra fluid is placed subcutaneously.
  Interventions: Other: Saline infiltration

INTERVENTIONS:
Drug: Exparel — liposomal bupivacaine wound infiltration
  Other Names: liposomal bupivacaine
  Arms: liposomal bupivacaine infiltration
Other: Saline infiltration — saline wound infiltration
  Arms: Saline infiltration

SUMMARY:
The aim of this study is to determine if local wound infiltration with liposomal bupivacaine at the time of cesarean delivery can decrease opioid use and provide adequate post-operative pain control.

DETAILED DESCRIPTION:
Specific Aim 1: To identify the effect of local infiltration of all wound layers with liposomal bupivacaine on opioid consumption up to 48 hours after cesarean delivery.

For this aim, in-patient narcotic use, measured in morphine equivalents, will be documented by the nurses and totaled during each 24 hour period after cesarean section until discharge.

Specific Aim 2: To identify the effect of local infiltration of all wound layers with liposomal bupivacaine on other, relevant, clinical outcomes, including time to first opiate use, time to mobility, occurrence of vomiting, use of rescue antiemetic medications, pain scores, and use of additional measures for pain control such as heating pads, muscle relaxers, gabapentin, between the study groups.

Specific Aim 3: To determine the occurrence of adverse events in the infants of breastfeeding women who have received local infiltration of all wound layers with liposomal bupivacaine compared to breastfeeding women who received saline infiltration.

Study Methods:

Patients will be randomized to either receive 20 mL liposomal bupivacaine diluted to 90 mL (treatment group), or 90 mL normal saline (control group). Patients with a BMI greater than or equal to 40 will receive 150 mL normal saline of the liposomal bupivacaine formulation. Randomization will occur in a 1:1 fashion via Miami Valley Pharmacy staff. All patients will be given the current medications used during cesarean delivery at MVH including Duramorph in the spinal or epidural via the Anesthesia team, Toradol for 24 hours on scheduled followed by Motrin on schedule until discharge.

Instillation of the liposomal bupivacaine or saline will be performed by resident physicians supervised by Wright State or private attending physicians. For each study group, 45 mL of their given solution will be infiltrated into the sub-fascial layer after its closure. Using an 18-gauge needle, 10 mL aliquots will be instilled into each lateral edge and six 2-mL aliquots into the superior and inferior fascial edges.

Post-operative care will first take place in the PACU in the usual fashion according to the anesthesiologist. The anesthesiologists will be blinded to the study group and patients will be given rescue parenteral opioids as deemed necessary.

The primary outcome of this study will be total oral morphine equivalents at 48 hours from the time of surgery. Nurses blind to the study group will record the total amount of opioid medications each patient used. This will be converted to a morphine equivalent of 1mg oral oxycodone to 1.5mg oral morphine.

Selection of Patients:

Recruitment: Patients will be recruited from Miami Valley Hospital Labor and Delivery and from Five Rivers Center for Women's Health. Investigators will identify potential patients from those who are admitted to Labor and Delivery for a scheduled cesarean delivery. Investigators will explain the study to potential patients and will obtain written informed consent from patients who agree to participate in the study.

Data Management Data required for the study will be recorded in the medical record by physicians and nursing staff. Physicians will document the procedure for infiltration in operative notes, indicating that the patient was randomized to "active medication (Experel ®) or saline." MVH Pharmacy staff will record the randomization/treatment key. Investigators, nursing staff, and patients will be blinded to the medication given. Documentation of pain scores, opioid medications used, other pain control methods used (heating pads, muscle relaxers, gabapentin, etc.) will be done by the physicians and nursing staff according to standard procedures. Data collection will consist of medical record review to record data on the paper data collection forms.

Confidentiality of Data PHI will be limited to information needed for the study objectives. Patients will be assigned a study ID number on the paper data collection forms and in the spreadsheet. Patient name and MRN will be kept in a separate key that will allow re-identification only if necessary to complete data collection.

Risks:

There is a risk of a breach of confidentiality. Risks to the Mother: Liposomal bupivacaine (Exparel ®). Liposomal bupivacaine is FDA approved for use via wound infiltration for post-surgical pain control. The most common adverse events include nausea, constipation, and vomiting. There have been reports of adverse neurologic reactions with the use of local anesthetics. These include persistent anesthesia and paresthesia. CNS reactions are characterized by excitation and/or depression. Toxic blood concentrations depress cardiac conductivity and excitability which may lead to dysrhythmias, sometimes leading to death. Allergic-type reactions (e.g., anaphylaxis and angioedema) are rare and may occur as a result of hypersensitivity to the local anesthetic or to other formulation ingredients. There have been reports of chondrolysis (mostly in the shoulder joint) following intra-articular infusion of local anesthetics, which is an unapproved use. Cases of methemoglobinemia have been reported with local anesthetic use. 12 In a Cochrane Review of 20 studies that used local anesthetic wound infiltration after cesarean delivery, no adverse cardiovascular or central nervous system reactions were noted in any of the included studies. 9

Risks to the Infant: Liposomal bupivacaine is contraindicated in pregnant women. Therefore, the use of this medication will occur after the fetus is delivered. Liposomal bupivacaine and its metabolite, pipecoloxylidide, are noted to be present in breastmilk in small amounts. There is no available information on effects of the drug in the breastfed infant or effects of the drug on milk production. The Infant Risk Center has indicated that it is highly unlikely for plasma levels in the infant to reach a toxic level due to any exposure from breastmilk and suggests that use of liposomal bupivacaine is probably compatible with breastfeeding without restriction. 3

Potential Benefits: Patients may receive benefit from the study by experiencing better postoperative pain control or by reducing opiate medication use while maintaining acceptable pain control. The potential benefit to women in the future is to have an effective option for pain control after cesarean delivery that does not require opiate medications.

Statistical Considerations: Based on a previous study performed at this institution in a similar patient population the investigators anticipate a 25% reduction in total oral morphine equivalents at 48 hours. Using a power of 0.80 and an alpha of 0.05 the investigators will need 54 patients per group, or a total of 108 patients in order to detect a difference of this size.

Data Analysis: Analysis of the data will be performed by members of the investigative team using SPSS. Repeated measures ANOVA will be used to compare pain pill (non-opioid) use, opioid pain pill use (in morphine equivalents) and pain scores over time for the study groups. Additional post hoc t-tests will be used as needed to identify specific group differences at the individual time points as appropriate. Potential covariates including parity, previous cesarean delivery, previous surgical history, and BMI will be examined for impact on opioid pain pill use and pain scores. Frequencies for adverse events in infants will be used to identify the occurrence of adverse events in infants exposed to liposomal bupivacaine versus those not exposed (including those who were not breastfed and those who were breastfed among mothers receiving the saline infiltration).

ELIGIBILITY:
Inclusion Criteria:

* Are between 18 and 45 years of age, inclusive.
* Are undergoing a planned, primary or repeat, cesarean delivery without permanent sterilization.
* Have a BMI ≤ 60.
* Are able to read and understand English.

Exclusion Criteria:

* Have pre-eclampsia with severe features.
* Has been taking medication assisted treatment for opioid addiction during this pregnancy.
* Have known sensitivity to local anesthetic.
* Have a known sensitivity to non-steroidal anti-inflammatory medications.
* Planning to have a tubal ligation after the cesarean delivery.
* Are unable to receive neuraxial analgesia and/or Duramorph, a morphine formulation that is the standard of care for intrathecal anesthesia at MVH.
* Are prisoners.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women delivering by scheduled cesarean delivery
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Opioid (narcotic medication) use | at the end of 48 hours after delivery
  total opioid use, as morphine equivalents; sum of narcotic pain medications over 48 hours reported in morphine equivalents, by the Ohio Automated RX reporting system calculator, where hydrocodone 5 mg is 5 morphine equivalent dose (MED) and percocet 5 is 7.5 MED

SECONDARY OUTCOMES:
Average pain scores Day 1 | at the end of 24 hours after delivery
  Patient reported pain scores (0-10 where ten is the highest possible and 0 is no pain) as recorded by nursing staff, average post delivery in recovery and up to 23 hours and 59 minutes.
Average pain scores Day 2 | at the end of 48 hours after delivery
  Patient reported pain scores (0-10 where ten is the highest possible and 0 is no pain) as recorded by nursing staff, average from 24 hours to 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Kindig, DO, Principal Investigator — Wright State University
Locations (1):
- Miami Valley Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared on a case by case basis.

REFERENCES:
- [Background] Bamigboye AA, Hofmeyr GJ. Local anaesthetic wound infiltration and abdominal nerves block during caesarean section for postoperative pain relief. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006954. doi: 10.1002/14651858.CD006954.pub2. PMID 19588413
- [Background] Bamigboye AA, Justus HG. Ropivacaine abdominal wound infiltration and peritoneal spraying at cesarean delivery for preemptive analgesia. Int J Gynaecol Obstet. 2008 Aug;102(2):160-4. doi: 10.1016/j.ijgo.2008.03.019. Epub 2008 Jun 9. PMID 18538773
- [Background] Gasanova I, Alexander J, Ogunnaike B, Hamid C, Rogers D, Minhajuddin A, Joshi GP. Transversus Abdominis Plane Block Versus Surgical Site Infiltration for Pain Management After Open Total Abdominal Hysterectomy. Anesth Analg. 2015 Nov;121(5):1383-8. doi: 10.1213/ANE.0000000000000909. PMID 26252171
- [Background] Kalogera E, Bakkum-Gamez JN, Weaver AL, Moriarty JP, Borah BJ, Langstraat CL, Jankowski CJ, Lovely JK, Cliby WA, Dowdy SC. Abdominal Incision Injection of Liposomal Bupivacaine and Opioid Use After Laparotomy for Gynecologic Malignancies. Obstet Gynecol. 2016 Nov;128(5):1009-1017. doi: 10.1097/AOG.0000000000001719. PMID 27741199
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Sammour T, Kahokehr A, Soop M, Hill AG. Peritoneal damage: the inflammatory response and clinical implications of the neuro-immuno-humoral axis. World J Surg. 2010 Apr;34(4):704-20. doi: 10.1007/s00268-009-0382-y. PMID 20049432
- [Background] Yaklic JL; Maxwell RA; Urschel K; Robinson S; Dearmond MK; Lindheim SR Effect of Continuous Local Anesthetic Use for Pain Control and Narcotic Use After Cesarean Section: A Randomized Trial. Open J Surg. 2017; 1(1): 026-030
- [Background] State of Ohio Board of Pharmacy 2019. OARRS Rules Update - Spring 2019; Rules Update - Drug Distributors - Spring 2019; Rules Update - Terminal Distributors - Spring 2019; 2018. 2nd and 3rd Quarter - Rule Update pharmacy.ohio.gov